CLINICAL TRIAL: NCT07271563
Title: Assessment of Pentraxin Levels in the Gingival Fluid of Abutment Teeth in the Context of the Use of Fixed Dentures
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Andrzej Gala, Dr, Jagiellonian University
Other Study IDs: 1072.6120.131.2023
Record Dates: First submitted 2025-11-15; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Periodontal Disease; Periodontal Diseases; Prosthodontics
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Pentraxine test — Diagnostic test - in order to measure Pantraxine level in gingival fluid was performed.

SUMMARY:
The use of fixed dentures in prosthetic treatment requires a thorough analysis of clinical factors such as: the condition of the abutments subject to grinding procedures, the degree of their loosening, the extent of missing teeth, and the condition of the periodontal tissues. An important step in prosthetic treatment is planning subsequent procedures, including the grinding of the crowns of the natural teeth. Often, the initial stages of gingivitis are not visible during a clinical examination [1-4].

ELIGIBILITY:
Inclusion Criteria:

* appropriate age range of patients, indication for the use of fixed dentures, no signs of gingivitis in the clinical examination

Exclusion Criteria:

* any autoimmune disease or other systemic disease which could alter the course of periodontal disease, the desire to withdraw from participation in the research and the occurrence of general and local diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study material consist of 90 patients, of both sexes, aged between 35-48 years, who report for prosthetic treatment with fixed dentures to the University Dental Clinic at the Institute of Dentistry in Krakow, in the period: March 2023- August 2024.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Concentration of pentraxine | March 2023- August 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Institute, Krakow, Poland